CLINICAL TRIAL: NCT06396949
Title: The Relationship Between Diaphragm Muscle Thickness and Anxiety, Depression and Activities of Daily Living in Fibromyalgia Patients
Brief Title: The Relationship Between Diaphragm Muscle Thickness and Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 97
Record Dates: First submitted 2024-01-11; First posted 2024-05-02 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia; Anxiety; Depression; Diaphragm Issues
Keywords: Diaphragm thickness; Activities of daily living
MeSH Terms: conditions — Fibromyalgia; Anxiety Disorders; Depression | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Volunteer men and women diagnosed with fibromyalgia to ACR (American College of Rheumatology) 2016 criteria between the ages of 18 and 50 who applied to our clinic will be included in our study
  Interventions: Diagnostic Test: Fibromyalgia study form; Diagnostic Test: Pulmonary function test; Diagnostic Test: Ultrasonographic Diaphragm Thickness Measurement
- Control group: Healthy,volunteer men and women between the ages of 18-50 who applied to our clinic will be included in our study
  Interventions: Diagnostic Test: Fibromyalgia study form; Diagnostic Test: Pulmonary function test; Diagnostic Test: Ultrasonographic Diaphragm Thickness Measurement

INTERVENTIONS:
Diagnostic Test: Fibromyalgia study form — Fibromyalgia study form, consisting of clinical measurement, Fibromyalgia impact questionnaire (FIQ), Beck Anxiety Questionnaire and Beck Depression Questionnaire, Short-Form (SF)-36, who applied to the outpatient clinic with fibromyalgia will be filled in detail.
Diagnostic Test: Pulmonary function test — Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange. This information can help your healthcare provider diagnose and decide the treatment of certain lung disorders.
  The investigators will use handheld spirometry device for measurement. Three measurements will be made. In these three measurements; FEV1(Forced Expiratory Volume In One Second)(L), FEV1 (%predicted), FVC (Forced Vital Capacity) (L), FVC (%predicted), FEV1/FVC (%) and FEV1/FVC (%predicted) will be evaluated. The arithmetic average of the results of these three measurements will be taken.
  Other Names: Spirometry function test
Diagnostic Test: Ultrasonographic Diaphragm Thickness Measurement — Diaphragm thickness (millimeter-mm) will be measured in the supine position with a 6-14 Mhz lineer, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD.,P.R. China) at the end of inspiration and expiration from the intercostal space on the anterior axillary line. The measurements will be evaluated by making three measurements from the right 8-9. intercostal space where the diaphragm is best visualized. End-expiratory (Forced residual capacity-FRC) (millimeter-mm), end-inspiratory (Total Lung Capacity) (millimeter-mm) and thickening rate (%) (thickness TLC / thickness FRC) will be evaluated three times and the arithmetic average of these three measurements will be taken.

SUMMARY:
Fibromyalgia syndrome is characterized by chronic pain, fatigue, sleep problems and functional symptoms. Fatigue, anxiety and depression disorders, poor quality of life, sleep disorders, decreased concentration, and impaired cognitive functions are non-specific pain-related symptoms.

Various studies have reported decreased chest expansion, maximal ventilatory volume and maximal expiratory pressure in fibromyalgia patients with widespread body pain. Additionally, dyspnea is a symptom associated with respiratory muscle weakness and is associated with general fatigue. In these individuals, lower data are obtained in daily living activities and general health evaluation surveys. We did not find any study in the literature regarding the relationship between diaphragm thickness and fibromyalgia symptoms. In the light of these data, we aimed to evaluate the thickness of the diaphragm, one of the most important inspiratory muscles, in fibromyalgia patients.

DETAILED DESCRIPTION:
Demographic information of all individuals included in the study will be collected. Daily living activity will be evaluated with Short Form-36 (SF-36), Fibromyalgia Impact Questionnaire (FIQ), Pittsburgh Sleep Quality Questionnaire (PSQI) and Beck Depression Inventory. In order to evaluate the respiratory function test in both the fibromyalgia and control groups, three consecutive measurements will be taken with a hand spirometer and the arithmetic average of these three measurements will be recorded. In fibromyalgia and control patients, diaphragm thickness was measured at 8-9 degrees on the right anterior axillary line with a 6-14 Mhz linear, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD., P.R. China) in the supine position. It will be measured at the end of inspiration and expiration from the intercostal space. Three measurements will be made and the arithmetic average will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with fibromyalgia according to the 2016 ACR (American College of Rheumatology) diagnostic criteria without any comorbidities (such as liver, kidney failure, DM, rheumatic disease)
* Patients who underwent Pulmonary Function Test (PFT)
* Patients without pulmonary disease
* 18 -50 years old women and men

Exclusion Criteria:

* Congenital spinal, costal and diaphragmatic anomalies neuromuscular disease
* Respiratory system diseases that affect lung functions
* Patients who cannot cooperate with spirometry.
* Having surgery to the chest wall or spine
* Those with BMI > 25
* Those with liver, kidney failure, DM, rheumatic disease, neurological disease
* Individuals < 18 years and > 50 years old

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: It will consist of participants with fibromyalgia patients, according to the 2016 ACR (American College of Rheumatology) diagnostic criteria, who apply to the Physical Medicine and Rehabilitation Clinic of the University of Health Sciences Gaziosmanpasa Training and Research Hospital within the study date ranges, meet the inclusion and exclusion criteria and voluntarily agree to participate in the research. Healthy individuals identical in age and gender will be included in the study as a control group. Demographic information (Fibromyalgia study form, consisting of clinical measurement, Fibromyalgia impact questionnaire (FIQ), Beck Anxiety Questionnaire and Beck Depression Questionnaire, Short-Form (SF)-36, ) of all individuals involved in the recruitment will be collected.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia study form | Within 1 month of applying to the outpatient clinic
  Fibromyalgia study form, consisting of clinical measurement (2016 ACR (American College of Rheumatology) fibromyalgia diagnostic criteria, Fibromyalgia impact questionnaire (FIQ), Beck Anxiety Questionnaire and Beck Depression Questionnaire, Short-Form (SF)-36), who applied to the outpatient clinic with fibromyalgia will be filled in detail.
Pulmonary function test | Within 1 month of applying to the outpatient clinic
  The investigators will use handheld spirometry device for measurement. Three measurements will be made. In these three measurements; FEV1(Forced Expiratory Volume In One Second)(L), FEV1 (%predicted), FVC (Forced Vital Capacity) (L), FVC (%predicted), FEV1/FVC (%) and FEV1/FVC (%predicted) will be evaluated. The arithmetic average of the results of these three measurements will be taken.
Ultrasonographic Diaphragm Thickness Measurement | Within 1 month of applying to the outpatient clinic
  Diaphragm thickness (millimeter-mm) will be measured in the supine position with a 6-14 Mhz lineer, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD.,P.R. China) at the end of inspiration and expiration from the intercostal space on the anterior axillary line. The measurements will be evaluated by making three measurements from the right 8-9. intercostal space where the diaphragm is best visualized. End-expiratory (Forced residual capacity-FRC) (millimeter-mm), end-inspiratory (Total Lung Capacity) (millimeter-mm) and thickening rate (%) (thickness TLC / thickness FRC) (percentage) will be evaluated three times and the arithmetic average of these three measurements will be taken.
Fibromyalgia diagnostic criteria | Within 1 month of applying to the outpatient clinic
  2016 revised American College of Rheumatology fibromyalgia diagnostic criteria; A patient satisfies the modified 2016 fibromyalgia criteria if the following three conditions are met:
  1. Widespread pain index (WPI) ≥7 and symptom severity scale (SSS) score ≥5, or WPI of 4∼6 and SSS score ≥9. 2. Generalized pain, defined as pain in at least four of five regions, must be present. Jaw, chest, and abdominal pain are excluded from the generalized pain definition. 3. Symptoms have been generally present for at least 3 months. 4. A diagnosis of fibromyalgia is valid irrespective of other diagnoses. A diagnosis of fibromyalgia does not exclude the presence of other clinically important illnesses.
Fibromyalgia diagnostic criteria-Widespread pain index (WPI) | Within 1 month of applying to the outpatient clinic
  Ascertainment
  1. WPI: note the number of areas in which the patient has had pain over the past week. In how many areas has the patient had pain? Score will be between 0 and 19 (Region 1) (Left upper region); jaw, left shoulder girdle, left upper arm, left lower arm, (Region 2) (Right upper region); jaw, right shoulder girdle, right upper arm, right lower arm, (Region 3) (Left lower region); hip (buttock, trochanter), left upper leg, left lower leg, (Region 4) (Right lower region); hip (buttock, trochanter), right upper leg, right lower leg and (Region 5) (Axial region); neck, upper back, lower back, chest, abdomen
Fibromyalgia diagnostic criteria-Symptom severity scale (SSS) | Within 1 month of applying to the outpatient clinic
  2. SSS score Fatigue Waking unrefreshed Cognitive symptoms For each of the three symptoms above, indicate the level of severity over the past week using the following scale: 0=no problem 1=slight or mild problems, generally mild or intermittent 2=moderate, considerable problems, often present and/or at a moderate level 3=severe: pervasive, continuous, life-disturbing problems The SSS score is the sum of the severity scores of the three symptoms (fatigue, waking unrefreshed, and cognitive symptoms) (0∼9), plus the sum (0∼3) of the number of the following symptoms the patient has been bothered by that occurred during the previous 6 months: 1.Headaches (0∼1) 2. Pain or cramps in lower abdomen (0∼1) 3. Depression (0∼1). The final symptom severity score is between 0 and 12 The fibromyalgia severity scale is the sum of the WPI and SSS

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | Within 1 month of applying to the outpatient clinic
  The FIQ is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes. The FIQ is composed of 10 items. The first item contains 11 questions related to physical functioning - each question is rated on a 4 point Likert type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. Items 4 through 10 are horizontal linear scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression. The FIQ is scored in such a way that a higher score indicates a greater impact of the syndrome on the person. Thus the maximum possible score is 100. The average FM patient scores about 50, severely afflicted patients are usually 70 plus.
Beck Anxiety Inventory | Within 1 month of applying to the outpatient clinic
  The BAI is a rating scale used to evaluate the severity of anxiety symptoms. The scale was developed by Aaron T Beck, MD.The BAI contains 21 self-report items. The items reflect symptoms of anxiety, including: numbness or tingling, feeling hot, wobbliness in legs, ability to relax, fear of the worst happening, dizziness or lightheadedness, pounding or racing heart, unsteadiness, feeling terrified, feeling nervous, feeling of choking, hands trembling, feeling shaky, fear of losing control, difficulty breathing, fear of dying, feeling scared, indigestion or abdominal discomfort, faintness, face flushing, and sweating. Each item allows the patient four choices from no symptom to severe symptom. For each item, the patient is asked to report how he or she has felt during the past week. The items are scored as 0, 1, 2, or 3. The score range is 0-63. A total score of 0-7 is considered minimal range, 8-15 is mild, 16-25 is moderate, and 26-63 is severe.
Beck Depression Inventory | Within 1 month of applying to the outpatient clinic
  The Beck Depression Inventory (BDI) is a 21-item, self-rated scale that evaluates key symptoms of depression including mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, suicidal ideas, crying, irritability, social withdrawal, indecisiveness, body image change, work difficulty, insomnia, fatigability, loss of appetite, weight loss, somatic preoccupation, and loss of libido. Individual scale items are scored on a 4-point continuum (0=least, 3=most), with a total summed score range of 0-63. Higher scores indicate greater depressive severity
Short Form- 36 (SF-36) | Within 1 month of applying to the outpatient clinic
  The SF-36 is a health status profile originally designed to measure health status of patients and outcomes of patients.The 36 questions on the SF-36 are meant to reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social function, emotional role, and mental health. The categories of physical role and emotional role reflect performance at the activity and participation levels.To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Ciftci, MD,Associate Professor, Principal Investigator — Kirklareli University Faculty of Health Sciences
Locations (1):
- Deniz Oke, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Result] Sarzi-Puttini P, Giorgi V, Atzeni F, Gorla R, Kosek E, Choy EH, Bazzichi L, Hauser W, Ablin JN, Aloush V, Buskila D, Amital H, Da Silva JAP, Perrot S, Morlion B, Polati E, Schweiger V, Coaccioli S, Varrassi G, Di Franco M, Torta R, Oien Forseth KM, Mannerkorpi K, Salaffi F, Di Carlo M, Cassisi G, Batticciotto A. Fibromyalgia position paper. Clin Exp Rheumatol. 2021 May-Jun;39 Suppl 130(3):186-193. doi: 10.55563/clinexprheumatol/i19pig. Epub 2021 May 13. PMID 34001303
- [Result] Alciati A, Nucera V, Masala IF, Giallanza M, La Corte L, Giorgi V, Sarzi-Puttini P, Atzeni F. One year in review 2021: fibromyalgia. Clin Exp Rheumatol. 2021 May-Jun;39 Suppl 130(3):3-12. doi: 10.55563/clinexprheumatol/gz4i3i. Epub 2021 May 13. PMID 34001307
- [Result] Ortiz-Rubio A, Torres-Sanchez I, Cabrera-Martos I, Lopez-Lopez L, Rodriguez-Torres J, Granados-Santiago M, Valenza MC. Respiratory disturbances in fibromyalgia: A systematic review and meta-analysis of case control studies. Expert Rev Respir Med. 2021 Sep;15(9):1217-1227. doi: 10.1080/17476348.2021.1918547. Epub 2021 Apr 26. PMID 33857393
- [Result] Tomas-Carus P, Biehl-Printes C, Del Pozo-Cruz J, Parraca JA, Folgado H, Perez-Sousa MA. Effects of respiratory muscle training on respiratory efficiency and health-related quality of life in sedentary women with fibromyalgia: a randomised controlled trial. Clin Exp Rheumatol. 2022 Jun;40(6):1119-1126. doi: 10.55563/clinexprheumatol/0v55nh. Epub 2022 Jun 22. PMID 35748715
- [Result] Noda Y, Sekiguchi K, Kohara N, Kanda F, Toda T. Ultrasonographic diaphragm thickness correlates with compound muscle action potential amplitude and forced vital capacity. Muscle Nerve. 2016 Apr;53(4):522-7. doi: 10.1002/mus.24902. Epub 2015 Oct 10. PMID 26357011